CLINICAL TRIAL: NCT03014037
Title: Comparing Mesenchymal Stem Cell Counts in Unilateral vs. Bilateral Posterior Superior Iliac Spine Bone Marrow Aspiration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Kenneth Mautner, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00093044
Record Dates: First submitted 2017-01-05; First posted 2017-01-09 (Estimated); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: Osteoarthritis
Keywords: Orthopedics
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unilateral Procurement of Bone Marrow (Other): Participants currently scheduled to undergo a bone marrow aspirate concentration (BMAC) procedure will be randomized to unilateral procurement of bone marrow.
  Interventions: Procedure: Unilateral Bone Marrow Procurement
- Bilateral Bone Marrow Procurement (Experimental): Participants currently scheduled to undergo a bone marrow aspirate concentration (BMAC) procedure will be randomized to bilateral procurement of bone marrow.
  Interventions: Procedure: Bilateral Bone Marrow Procurement

INTERVENTIONS:
Procedure: Unilateral Bone Marrow Procurement — A total of 61cc of bone marrow will be procured under ultrasound guidance from one posterior superior iliac spine (PSIS) via 3 passes, each at least 1 cm apart, through the bone cortex. In each pass, investigators will obtain 2.3cc of BMA with a 60cc syringes.
  Arms: Unilateral Procurement of Bone Marrow
Procedure: Bilateral Bone Marrow Procurement — 30.5cc of bone marrow will be obtained under ultrasound guidance from each posterior superior iliac spine (PSIS) with 3 passes, at least 1 cm apart, per side (10.17cc per pass) using 60cc syringes. The collection from each PSIS will be combined to yield a total of 61cc.
  Arms: Bilateral Bone Marrow Procurement

SUMMARY:
Musculoskeletal conditions are common sources of pain. Specifically, osteoarthritis affects nearly 27 million people in the United States. This disease leads to the breakdown of the cartilage surfaces of the joints, which serve as the connection points between the bones of the body, causing a large amount of pain and disability in patients. Increasing the number of available treatment options for osteoarthritis is becoming increasingly more important as Americans continue to age. Using stem cells taken from bone marrow is one of the non-operative treatments that has been gaining popularity in the recent past. This study aims to clarify how this procedure should best be done by comparing stem cell concentrations and patient outcomes (short and long term) in patients who have stem cells taken from one area vs two (unilateral vs bilateral posterior superior iliac spine (PSIS) aspirations).

DETAILED DESCRIPTION:
Musculoskeletal conditions are common sources of pain. Specifically, osteoarthritis affects nearly 27 million people in the United States. This disease leads to the breakdown of the cartilage surfaces of the joints, which serve as the connection points between the bones of the body, causing a large amount of pain and disability in patients. Increasing the number of available treatment options for osteoarthritis is becoming increasingly more important as Americans continue to age. Using stem cells taken from bone marrow is one of the non-operative treatments that has been gaining popularity in the recent past. This study aims to clarify how this procedure should best be done by comparing stem cell concentrations and patient outcomes (short and long term) in patients who have stem cells taken from one area vs two (unilateral vs bilateral posterior superior iliac spine (PSIS) aspirations).

This research study involves the participant being randomly placed into one of two groups; one group will have cells taken from one hip, and the other will have cells taken from both hips. Both of these approaches are performed in clinics currently, and both are considered to be standard of care. All bone marrow collected for the purposes of this study will be obtained by the principal investigator while performing the standard procedure. In obtaining these sample the physicians will abide by the standard of care set forth for the Bone Marrow Aspiration Concentrate procedure.

ELIGIBILITY:
Inclusion Criteria:

* Currently scheduled for a bone marrow aspirate concentration (BMAC) procedure
* Cognitively able to give consent and complete the required questionnaires

Exclusion Criteria:

* History of leukemia or lymphoma
* History of any autoimmune disorders and disease
* Currently taking immunosuppressive medications
* Presence of an active or suspected infection, or an infection of the joint in question within the past 6 months
* Vulnerable populations (pregnant women and breast-feeding women)
* Cortisone injection into the affected joint within 6 weeks
* Used NSAIDs within 1 week of the procedure
* History of bleeding disorders or inflammatory joint disease
* Surgical intervention on the affected or contralateral joint within 6 months of BMAC injection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-09-07 (Actual); Primary Completion 2020-06-13 (Actual); Study Completion 2020-06-13 (Actual)

PRIMARY OUTCOMES:
Change Quality of Life assessed by the Emory Quality of Life (EQOL) Survey Score | Pre-treatment, Follow Up (Up to One Year)
  The EQOL survey measures five dimensions - mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The participant will be asked to answer questions regarding these measures and to indicate their current experience on a scale from 1 to 3; 1 being "no problem" and 3 being "most extreme problem". The answers to these question are put together to create a 5 digit composite score.This composite score can be indexed to a lookup table which produces a single summary score from 0 to 100. The lookup table we use is weighted and normalized to the United Stated general population.
Change in the Knee Injury and Osteoarthritis Outcome Score (KOOS) | Pre-treatment, Follow Up (Up to One Year)
  The KOOS questionnaire is an instrument to assess the patient's opinion about their osteoarthritis and associated problems. It consists of 5 subscales; Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of life (QOL). Standardized answer options are given (5 Likert boxes) and each question is assigned a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale. A total lower score indicates more problems.

SECONDARY OUTCOMES:
Capacity of Isolated Cells to Differentiate Down Cell Lineages | Post Cell Culture (Up to 21 Days)
  Bone marrow aspirate will be placed in 10 mL heparinized tubes and nucleated cells will be isolated with a density gradient and re-suspended in complete culture medium for plating. Isolated adherent cells will be processed for the ability to differentiate down osteogenic-, adipogenic- and chondrogenic-lineage after cell harvest. Specifically, isolated cells are treated with different media to induce their differentiation into 1) osteo-progenitor cells (identified by positive staining with Alzarian red, 2) adipocytes (identified by positive staining with Oil-Red) and 3) chondrocytes (identified by positive staining with Alcian blue). The presence of these phenotypes should be prevalent by 3 weeks; if not, the cells are not considered pluripotent for that lineage and hence would not be classified as mesenchymal stem cells.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Mautner, MD, Principal Investigator — Emory University
Locations (1):
- The Emory Clinic, Atlanta, Georgia, United States